CLINICAL TRIAL: NCT04594369
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of Brensocatib Administered Once Daily for 52 Weeks in Subjects With Non-Cystic Fibrosis Bronchiectasis - The ASPEN Study
Brief Title: A Study to Assess the Efficacy, Safety, and Tolerability of Brensocatib in Participants With Non-Cystic Fibrosis Bronchiectasis
Acronym: ASPEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS1007-301; 2020-003688-25 (EudraCT Number)
Expanded Access: NCT05344508 (Approved for marketing)
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Non-Cystic Fibrosis Bronchiectasis
Keywords: ASPEN; Brensocatib; INS1007
MeSH Terms: interventions — brensocatib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brensocatib 10 milligrams (mg) (Experimental): Participants will receive brensocatib 10 mg, tablets orally, once daily, for 52 weeks.
  Interventions: Drug: Brensocatib 10 mg
- Brensocatib 25 mg (Experimental): Participants will receive brensocatib 25 mg, tablets orally, once daily, for 52 weeks.
  Interventions: Drug: Brensocatib 25 mg
- Placebo (Placebo Comparator): Participants will receive a brensocatib-matching placebo, tablets orally, once daily, for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brensocatib 10 mg — Oral tablet.
  Other Names: INS1007
  Arms: Brensocatib 10 milligrams (mg)
Drug: Brensocatib 25 mg — Oral tablet.
  Other Names: INS1007
  Arms: Brensocatib 25 mg
Drug: Placebo — Brensocatib-matching oral tablet.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of brensocatib at 10 mg and 25 mg compared with placebo on the rate of pulmonary exacerbations (PEs) over the 52-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Provide their signed study informed consent to participate.

   a. Adolescent participants must have signed study assent form to participate, and the adolescent's parent or legal guardian must have provided signed informed consent for the adolescent to participate.
2. Clinical history consistent with non-cystic fibrosis bronchiectasis (NCFBE) (cough, chronic sputum production and/or recurrent respiratory infections) that is confirmed by chest computerized tomography (CT) scan.
3. At least 2 PEs defined by need for antibiotic prescription by a physician for the signs and symptoms of respiratory infections in the past 12 months before the Screening Visit.

   a. Adolescent participants are required to have at least 1 pulmonary exacerbation in the prior 12 months.
4. Women must be postmenopausal (defined as no menses for 12 months without an alternative medical cause), surgically sterile, or using highly effective contraception (ie, methods that can achieve a failure rate <1% per year when used consistently and correctly) from Day 1 to at least 90 days after the last dose.
5. Male participants with female partners of childbearing potential must be using effective contraception from Day 1 to at least 90 days after the last dose.
6. Male participants with pregnant or non-pregnant women of child-bearing potential partners must use condoms to avoid potential exposure to the embryo/fetus.

Exclusion Criteria:

1. A primary diagnosis of chronic obstructive pulmonary disease (COPD) or asthma as judged by the Investigator.
2. Bronchiectasis due to cystic fibrosis.
3. Current smokers as defined per Centers for Disease Control (CDC).
4. Known or suspected immunodeficiency disorder, including history of invasive opportunistic infections.
5. Known history of human immunodeficiency virus (HIV) infection.
6. Currently being treated for nontuberculous mycobacteria (NTM) lung infection, allergic bronchopulmonary aspergillosis, or tuberculosis (TB).
7. Active and current symptomatic infection by 2019 corona virus disease (COVID-19).
8. Inability to follow the procedures of the study (eg, due to language problems or psychological disorders).
9. Receiving medications or therapy that are prohibited as concomitant medications.
10. Previously participated in a clinical trial for brensocatib.
11. Received any live attenuated vaccine within 4 weeks prior to the first administration of brensocatib.
12. Suffering an exacerbation 4 weeks before Screening or during the Screening period.
13. Adult participants only: Have compliance issues with completion of electronic diary entries during the Screening Period and in the opinion of the Investigator, compliance is unlikely to improve during the study.
14. Participated in any other interventional clinical studies within 3 months before Screening Visit.
15. History of alcohol or drug abuse within 6 months prior to the Screening Visit.
16. Is the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.
17. Known history of hypersensitivity to brensocatib or any of its excipients.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1767 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (373):
- United States (67):
  - USA013, Birmingham, Alabama
  - USA080, Conway, Arkansas
  - USA044, Little Rock, Arkansas
  - USA104, Fresno, California
  - USA055, Los Angeles, California
  - USA029, Newport Beach, California
  - USA102, Northridge, California
  - USA022, Palm Springs, California
  - USA024, Sacramento, California
  - USA035, San Diego, California
  - USA078, Santa Barbara, California
  - USA027, Ventura, California
  - USA075, Denver, Colorado
  - USA017, Farmington, Connecticut
  - USA001, Washington D.C., District of Columbia
  - USA015, Clearwater, Florida
  - USA076, Gainesville, Florida
  - USA082, Jacksonville, Florida
  - USA039, Kissimmee, Florida
  - USA072, Leesburg, Florida
  - USA037, Miami, Florida
  - USA019, Miami Lakes, Florida
  - USA049, Naples, Florida
  - USA052, Orlando, Florida
  - USA103, Plantation, Florida
  - USA084, Sarasota, Florida
  - USA089, St. Petersburg, Florida
  - USA074, St. Petersburg, Florida
  - USA120, Tampa, Florida
  - USA012, Atlanta, Georgia
  - USA053, Augusta, Georgia
  - USA073, Chicago, Illinois
  - USA061, Maywood, Illinois
  - USA115, Hammond, Indiana
  - USA063, Iowa City, Iowa
  - USA031, Kansas City, Kansas
  - USA020, New Orleans, Louisiana
  - USA051, New Orleans, Louisiana
  - USA003, Baltimore, Maryland
  - USA079, Boston, Massachusetts
  - USA064, Springfield, Massachusetts
  - USA010, Rochester, Minnesota
  - USA006, Chesterfield, Missouri
  - USA059, St Louis, Missouri
  - USA110, Lincoln, Nebraska
  - USA065, Toms River, New Jersey
  - USA066, New Hyde Park, New York
  - USA021, New York, New York
  - USA085, New York, New York
  - USA033, Gastonia, North Carolina
  - USA096, Huntersville, North Carolina
  - USA026, Winston-Salem, North Carolina
  - USA067, Cincinnati, Ohio
  - USA093, Cleveland, Ohio
  - USA023, Portland, Oregon
  - USA038, DuBois, Pennsylvania
  - USA046, Philadelphia, Pennsylvania
  - USA005, Charleston, South Carolina
  - USA036, Rock Hill, South Carolina
  - USA041, Franklin, Tennessee
  - USA109, Nashville, Tennessee
  - USA097, Dallas, Texas
  - USA050, McKinney, Texas
  - USA011, San Antonio, Texas
  - USA002, Tyler, Texas
  - USA034, Williamsburg, Virginia
  - USA088, Vancouver, Washington
- Argentina (23):
  - ARG027, Bahía Blanca, Buenos Aires
  - ARG021, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - ARG022, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - ARG002, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - ARG001, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - ARG003, Ciudad Autónoma de BuenosAires, Buenos Aires
  - ARG004, Ciudad Autónoma de BuenosAires, Buenos Aires
  - ARG006, La Plata, Buenos Aires
  - ARG013, Mar del Plata, Buenos Aires
  - ARG017, Mar del Plata, Buenos Aires
  - ARG009, Villa Vatteone, Buenos Aires
  - ARG012, Buenos Aires, Ciudad Autónoma de BuenosAires
  - ARG018, Buenos Aires, Ciudad Autónoma de BuenosAires
  - ARG026, Recoleta, Ciudad Autónoma de BuenosAires
  - ARG023, Río Cuarto, Córdoba Province
  - ARG014, Vistalba, Mendoza Province
  - ARG010, Rosario, Santa Fe Province
  - ARG015, San Miguel de Tucumán, Tucumán Province
  - ARG025, San Miguel de Tucumán, Tucumán Province
  - ARG005, Córdoba
  - ARG007, Mendoza
  - ARG011, Rosario
  - ARG019, Santa Fe
- Australia (18):
  - AUS013, Kogarah, New South Wales
  - AUS008, New Lambton Heights, New South Wales
  - AUS007, Westmead, New South Wales
  - AUS012, Cairns North, Queensland
  - AUS001, Chermside, Queensland
  - AUS010, Greenslopes, Queensland
  - AUS006, South Brisbane, Queensland
  - AUS019, South Brisbane, Queensland
  - AUS011, Adelaide, South Australia
  - AUS017, Bedford Park, South Australia
  - AUS022, North Adelaide, South Australia
  - AUS009, Woodville South, South Australia
  - AUS002, Box Hill, Victoria
  - AUS014, Clayton, Victoria
  - AUS018, Murdoch, Western Australia
  - AUS005, Nedlands, Western Australia
  - AUS003, Concord
  - AUS015, Spearwood
- AUT002, Linz, Austria
- Belgium (7):
  - BEL002, Ghent, Oost-Vlaanderen
  - BEL009, Ghent, Oost-Vlaanderen
  - BEL004, Roeselare, West-Vlaanderen
  - BEL001, Leuven
  - BEL007, Liège
  - BEL003, Mechelen
  - BEL008, Sint-Niklaas
- Brazil (7):
  - BRA009, Passo Fundo, Rio Grande do Sul
  - BRA005, Porto Alegre, Rio Grande do Sul
  - BRA001, Blumenau, Santa Catarina
  - BRA006, Santo André, São Paulo
  - BRA003, Botucatu
  - BRA004, São Bernardo do Campo
  - BRA011, São Paulo
- Bulgaria (17):
  - BGR011, Sofia, Sofia-Grad
  - BGR009, Sofia, Sofia-Grad
  - BGR002, Sofia, Sofia-Grad
  - BGR005, Blagoevgrad
  - BGR006, Gabrovo
  - BGR014, Kozloduy
  - BGR015, Lovech
  - BGR007, Montana
  - BGR018, Pazardzhik
  - BGR019, Pleven
  - BGR004, Plovdiv
  - BGR008, Rousse
  - BGR017, Sliven
  - BGR010, Sofia
  - BGR012, Veliko Tarnovo
  - BGR013, Vidin
  - BGR016, Vratsa
- Canada (2):
  - CAN004, Toronto, Ontario
  - CAN002, Montreal, Quebec
- Chile (7):
  - CHL007, Valdivia, Los Ríos Region
  - CHL005, Curicó, Maule Region
  - CHL010, Talca, Maule Region
  - CHL001, Providencia, Región-MetropolitanadeSantiago
  - CHL002, Providencia, Región-MetropolitanadeSantiago
  - CHL008, Providencia, Región-MetropolitanadeSantiago
  - CHL004, Quillota
- Colombia (6):
  - COL001, Bogotá, Bogota D.C.
  - COL006, Zipaquirá, Cundinamarca
  - COL005, Floridablanca, Santander Department
  - COL003, Cali, Valle del Cauca Department
  - COL002, Bogota DC
  - COL004, Santiago de Cali
- Denmark (8):
  - DNK008, Copenhagen O, Capital
  - DNK001, Hvidovre, Capital
  - DNK005, Odense C, Region Syddanmark
  - DNK006, Vejle, Region Syddanmark
  - DNK003, Aalborg
  - DNK007, Aarhus
  - DNK004, Hellerup
  - DNK002, Roskilde
- France (8):
  - FRA002, Strasbourg, Bas-Rhin
  - FRA005, Montpellier, Hérault
  - FRA004, Amiens
  - FRA011, Créteil
  - FRA003, Nantes
  - FRA009, Nice
  - FRA010, Paris
  - FRA006, Toulouse
- Germany (19):
  - DEU009, Heidelberg, Baden-Wurttemberg
  - DEU025, München, Bavaria
  - DEU027, Potsdam, Brandenburg
  - DEU008, Frankfurt am Main, Hesse
  - DEU005, Marburg, Hesse
  - DEU031, Hanover, Lower Saxony
  - DEU013, Essen, North Rhine-Westphalia
  - DEU003, Leipzig, Saxony
  - DEU016, Halle, Saxony-Anhalt
  - DEU020, Geesthacht, Schleswig-Holstein
  - DEU002, Berlin
  - DEU019, Berlin
  - DEU006, Berlin
  - DEU011, Berlin
  - DEU014, Dresden
  - DEU021, Frankfurt
  - DEU015, Hanover
  - DEU023, Mainz
  - DEU029, Münster
- Greece (3):
  - GRC003, Alexandroupoli, Evros
  - GRC007, Heraklion
  - GRC006, Thessaloniki
- HUN005, Tatabánya, Komárom-Esztergom, Hungary
- Ireland (3):
  - IRL003, Dublin
  - IRL002, Dublin
  - IRL001, Limerick
- Israel (10):
  - ISR001, Ashkelon
  - ISR010, Beersheba
  - ISR008, Haifa
  - ISR006, Jerusalem
  - ISR002, Jerusalem
  - ISR009, Kefar Sava
  - ISR011, Petah Tikva
  - ISR007, Ramat Gan
  - ISR003, Rehovot
  - ISR004, Ẕerifin
- Italy (11):
  - ITA010, Bologna, Emilia-Romagna
  - ITA008, Ferrara, Emilia-Romagna
  - ITA002, Reggio Emilia, Emilia-Romagna
  - ITA006, Milan, Lombardy
  - ITA012, Milan, Lombardy
  - ITA011, Rozzano, Lombardy
  - ITA004, Siena, Tuscany
  - ITA003, Milan
  - ITA001, Palermo
  - ITA007, Pavia
  - ITA009, Roma
- Japan (29):
  - JPN029, Toyoake, Aiti
  - JPN031, Toon-Shi, Ehime
  - JPN027, Fukuoka, Hukuoka
  - JPN023, Iizuka-Shi, Hukuoka
  - JPN009, Kobe, Hyôgo
  - JPN020, Kasama-Shi, Ibaraki
  - JPN001, Naka-gun, Ibaraki
  - JPN022, Takamatsu, Kagawa-ken
  - JPN028, Yokohama-Shi Konan-Ku, Kanagawa
  - JPN005, Koshi Shi, Kumamoto
  - JPN008, Matsusaka-shi, Mie-ken
  - JPN011, Tsu, Mie-ken
  - JPN034, Sendai, Miyagi
  - JPN013, Nagasaki, Nagasaki
  - JPN012, Chuo-ku, Niigata
  - JPN015, Matsue, Shimane
  - JPN007, Kiyose, Tokyo
  - JPN014, Ōta-ku, Tokyo
  - JPN006, Shinagawa-ku, Tokyo
  - JPN017, Shinagawa-ku, Tokyo
  - JPN002, Shinjuku-ku, Tokyo
  - JPN032, Shinjuku-ku, Tokyo
  - JPN019, Shimonoseki-Shi, Yamaguchi
  - JPN030, Fukuoka
  - JPN003, Hamamatsu
  - JPN004, Kita Kyushu-shi
  - JPN016, Matsue
  - JPN010, Meguro-ku
  - JPN018, Toyonaka-shi
- Latvia (2):
  - LVA002, Daugavpils, Daugavpils Aprinkis
  - LVA005, Jūrmala
- Malaysia (4):
  - MYS004, Kuantan, Pahang
  - MYS001, Kuala Lumpur, WilayahPersekutuan KualaLumpur
  - MYS003, Kota Bharu
  - MYS005, Kuala Lumpur
- Mexico (8):
  - MEX007, Guadalajara, Jalisco
  - MEX008, Guadalajara, Jalisco
  - MEX005, Guadalajara, Jalisco
  - MEX004, Guadalajara, Jalisco
  - MEX003, Monterrey, Nuevo León
  - MEX006, Durango
  - MEX001, Monterrey
  - MEX002, Oaxaca City
- Netherlands (4):
  - NLD003, Arnhem, Gelderland
  - NLD001, Alkmaar, North Holland
  - NLD002, Amsterdam, North Holland
  - NLD006, Rotterdam
- New Zealand (10):
  - NZL006, Otahuhu, Auckland
  - NZL009, Hastings, Hawkes's Bay
  - NZL005, Christchurch, South Island
  - NZL001, Dunedin, South Island
  - NZL002, Hamilton, Waikato Region
  - NZL011, Paraparaumu, Wellington Region
  - NZL003, Auckland
  - NZL008, Auckland
  - NZL007, Tauranga
  - NZL010, Wellington
- Peru (5):
  - PER005, Chancay
  - PER001, Lima
  - PER003, Lima
  - PER002, Lima
  - PER006, Piura
- Poland (14):
  - POL005, Bialystok
  - POL006, Bielsko-Biala
  - POL016, Katowice
  - POL015, Kielce
  - POL017, Krakow
  - POL018, Ksawerów
  - POL008, Rabka-Zdrój
  - POL011, Rzeszów
  - POL010, Siedlce
  - POL007, Sosnowiec
  - POL001, Sucha Beskidzka
  - POL014, Szczecin
  - POL009, Tarnów
  - POL012, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Portugal (5):
  - PRT005, Aveiro
  - PRT009, Braga
  - PRT006, Guarda
  - PRT002, Guimarães
  - PRT003, Lisbon
- Serbia (5):
  - SRB001, Belgrade
  - SRB003, Belgrade
  - SRB007, Niš
  - SRB014, Sombor
  - SRB010, Užice
- Slovakia (2):
  - SVK002, Bardejov
  - SVK003, Spisská Nová Ves
- South Korea (11):
  - KOR015, Ansan-si, Gyeonggido
  - KOR008, Bucheon-si, Gyeonggido
  - KOR007, Seongnam-si, Gyeonggido
  - KOR003, Seoul, Seoul Teugbyeolsi
  - KOR004, Incheon
  - KOR012, Seoul
  - KOR011, Seoul
  - KOR009, Seoul
  - KOR013, Seoul
  - KOR010, Seoul
  - KOR005, Seoul
- Spain (12):
  - ESP009, Santiago de Compostela, A Coruña
  - ESP013, Badalona, Barcelona
  - ESP012, Santander, Cantabria
  - ESP015, Pozuelo de Alarcón, Madrid
  - ESP011, Pamplona, Navarre
  - ESP008, Oviedo, Principality of Asturias
  - ESP003, Barcelona
  - ESP016, Barcelona
  - ESP001, Girona
  - ESP006, L'Hospitalet de Llobregat
  - ESP007, Madrid
  - ESP002, Madrid
- Taiwan (7):
  - TWN003, Kaohsiung City
  - TWN002, Kaohsiung City
  - TWN001, Kaohsiung City
  - TWN005, New Taipei City
  - TWN007, Taipei
  - TWN004, Taipei
  - TWN006, Taipei
- Thailand (3):
  - THA004, Nakhonnayok, Changwat Nakhon Nayok
  - THA002, Muang, Changwat Nonthaburi
  - THA003, Khon Kaen
- Turkey (Türkiye) (9):
  - TUR006, Atakum, Samsun
  - TUR010, Ankara
  - TUR011, Ankara
  - TUR003, Çanakkale
  - TUR008, Izmir
  - TUR004, Izmir
  - TUR009, Kocaeli
  - TUR005, Konya
  - TUR001, Mersin
- Ukraine (9):
  - UKR001, Kharkiv, Kharkivs’ka Oblast’
  - UKR007, Kherson, Kherson Oblast
  - UKR005, Poltava, Poltava Oblast
  - UKR012, Dnipro
  - UKR009, Ivano-Frankivsk
  - UKR008, Kyiv
  - UKR004, Kyiv
  - UKR003, Odesa
  - UKR010, Vinnytsia
- United Kingdom (16):
  - GBR001, Cambridge, Cambridgeshire
  - GBR015, Exeter, Devon
  - GBR017, Norwich, Norfolk
  - GBR013, Llandough, Vale of Glamorgan, the
  - GBR016, Bradford, Yorkshire
  - GBR006, Birmingham
  - GBR002, Chertsey
  - GBR007, Dundee
  - GBR004, Liverpool
  - GBR009, London
  - GBR008, Manchester
  - GBR011, Manchester
  - GBR003, Newcastle upon Tyne
  - GBR012, Salford
  - GBR018, Southampton
  - GBR010, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morimoto K, Chalmers JD, Burgel PR, Daley CL, De Soyza A, Mauger D, Metersky ML, Zhang X, Li S, Goto Y, Teper A, Fernandez C, Hasegawa N. Efficacy and safety of brensocatib in Japanese patients with non-cystic fibrosis bronchiectasis: Analysis of the ASPEN trial. Respir Investig. 2026 Jan 9;64(2):101357. doi: 10.1016/j.resinv.2025.101357. Online ahead of print. PMID 41519018
- [Derived] Chalmers JD, Burgel PR, Daley CL, De Soyza A, Haworth CS, Mauger D, Loebinger MR, McShane PJ, Ringshausen FC, Blasi F, Shteinberg M, Mange K, Teper A, Fernandez C, Zambrano M, Fan C, Zhang X, Metersky ML; ASPEN Investigators. Phase 3 Trial of the DPP-1 Inhibitor Brensocatib in Bronchiectasis. N Engl J Med. 2025 Apr 24;392(16):1569-1581. doi: 10.1056/NEJMoa2411664. PMID 40267423
- [Derived] Chalmers JD, Burgel PR, Daley CL, De Soyza A, Haworth CS, Mauger D, Mange K, Teper A, Fernandez C, Conroy D, Metersky M. Brensocatib in non-cystic fibrosis bronchiectasis: ASPEN protocol and baseline characteristics. ERJ Open Res. 2024 Jul 22;10(4):00151-2024. doi: 10.1183/23120541.00151-2024. eCollection 2024 Jul. PMID 39040578
- [Derived] Chalmers JD, Usansky H, Rubino CM, Teper A, Fernandez C, Zou J, Mange KC. Pharmacokinetic/Pharmacodynamic Evaluation of the Dipeptidyl Peptidase 1 Inhibitor Brensocatib for Non-cystic Fibrosis Bronchiectasis. Clin Pharmacokinet. 2022 Oct;61(10):1457-1469. doi: 10.1007/s40262-022-01147-w. Epub 2022 Jul 25. PMID 35976570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 373 sites in 36 countries from 01 Dec 2020 to 28 Oct 2024.
Pre-assignment Details: A total of 2296 participants were screened, 1767 participants with non-cystic fibrosis bronchiectasis were enrolled in the study. Due to the war in Ukraine, 44 participants from Ukraine were discontinued and excluded from all analyses. There were 2 additional participants who were excluded from all analyses due to serious Good Clinical Practice (GCP) non-compliance. A total of 1721 participants were randomized and analyzed.
Groups:
- Brensocatib 10 Milligrams (mg): Participants received brensocatib 10 mg tablets, orally, once daily, for 52 weeks.
- Brensocatib 25 mg: Participants received brensocatib 25 mg tablets, orally, once daily, for 52 weeks.
- Placebo: Participants received a brensocatib matching placebo, tablets orally, once daily, for 52 weeks.
Period: Overall Study
Arm/Group | Brensocatib 10 Milligrams (mg) | Brensocatib 25 mg | Placebo
Started | 583 | 575 | 563
Completed | 458 | 466 | 457
Not Completed | 125 | 109 | 106
Not completed — Adverse Event | 10 | 10 | 9
Not completed — Death | 2 | 4 | 8
Not completed — Lost to Follow-up | 10 | 2 | 4
Not completed — Physician Decision | 2 | 2 | 3
Not completed — Protocol deviation | 1 | 3 | 2
Not completed — Withdrawal by Subject | 40 | 32 | 37
Not completed — Reason not specified | 60 | 56 | 43

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) analysis set included all participants who were randomized.
Groups:
- Brensocatib 10 mg: Participants received brensocatib 10 mg tablets, orally, once daily, for 52 weeks.
- Brensocatib 25 mg: Participants received brensocatib 25 mg tablets orally, once daily, for 52 weeks.
- Placebo: Participants received a brensocatib matching placebo tablets orally, once daily, for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo | Total
Number analyzed (Participants) | 583 | 575 | 563 | 1721
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (15.92) | 60.6 (15.78) | 60.0 (15.44) | 60.2 (15.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 385 | 360 | 362 | 1107
  Male | 198 | 215 | 201 | 614
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 177 | 164 | 170 | 511
  Not Hispanic or Latino | 391 | 397 | 373 | 1161
  Unknown or Not Reported | 15 | 14 | 20 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 8 | 6 | 9 | 23
  Race: Asian | 63 | 64 | 64 | 191
  Race: Black or African American | 2 | 5 | 3 | 10
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Race: White | 431 | 430 | 405 | 1266
  Race: Other | 15 | 13 | 11 | 39
  Race: Unknown or Not Reported | 48 | 46 | 59 | 153
  Race: More than one race | 15 | 11 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Pulmonary Exacerbations (PEs)
Description: PE was defined as having 3 or more of these symptoms for at least 48 hours resulting in a physician's decision to prescribe antibiotics: 1. Increased cough 2. Increased sputum volume or change in sputum consistency 3. Increased sputum purulence 4. Increased breathlessness and/or decreased exercise tolerance 5. Fatigue and/or malaise 6. Hemoptysis. A severe pulmonary exacerbation was that required intravenous (IV) antibacterial drug treatment and/or hospitalization. A minimum of 14 days must have occurred between one exacerbation onset and the next. Any exacerbation that occurred less than 14 days from the prior exacerbation was not considered a new exacerbation. Independent adjudication committee with pulmonary physicians adjudicated reported PE events to see if they fulfil the protocol definition. The rate of PE was analyzed using the negative binomial model.
Time Frame: Up to Week 52
Population: The ITT analysis set included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: exacerbation per participant-year
Groups:
- Brensocatib 10 mg: Participants received brensocatib 10 mg, tablets orally, once daily, for 52 weeks.
- Brensocatib 25 mg: Participants received brensocatib 25 mg, tablets orally, once daily, for 52 weeks.
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 583 | 575 | 563
exacerbation per participant-year | 1.015 [0.910 to 1.132] | 1.036 [0.927 to 1.157] | 1.286 [1.158 to 1.428]
Statistical Analysis 1: Comparison: Brensocatib 10 mg vs Placebo; Model treatment & randomization stratification factor=geographic region, sputum sample (Pseudomonas aeruginosa) at start & PE last 12 months, age group (fixed effects) & time at risk (log scale) as offset variable. Robust sandwich covariance estimator used; Test type: Superiority; p = 0.0019, Negative binomial regression — Adjusted p-value = 0.0038. The enhanced mixture-based gatekeeping procedure was used to control the overall type I error rate. Multiplicity adjusted p-value for the primary endpoint was tested at two-sided alpha = 0.01; Rate ratio = 0.789, 95% CI 2-sided [0.680 to 0.916]
Statistical Analysis 2: Comparison: Brensocatib 25 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0046, Negative binomial regression — Adjusted p-value = 0.0048. The enhanced mixture-based gatekeeping procedure was used to control the overall type I error rate. Multiplicity adjusted p-value for the primary endpoint was tested at two-sided alpha = 0.01; Rate ratio = 0.806, 95% CI 2-sided [0.694 to 0.936]

2. Secondary Outcome: Time to First PE
Description: PE was defined as having 3 or more of following symptoms for at least 48 hours resulting in physician's decision to prescribe antibiotics:1.Increased cough2.Increased sputum volume or change in sputum consistency3.Increased sputum purulence4.Increased breathlessness &/or decreased exercise tolerance5.Fatigue &/or malaise6.Hemoptysis.Severe PE were those requiring IV antibacterial drug treatment &/or hospitalization. Minimum of 14 days must have occurred between one exacerbation onset and next. Any exacerbation that occurred within 14 days of prior exacerbation was not considered a new exacerbation. Time to first PE was calculated from randomization date to onset date of the first exacerbation. Participants who did not have exacerbation at end of 52-week treatment period were considered as censored at date of Week 52 in Cox proportional hazard model. Independent adjudication committee with pulmonary physicians adjudicated reported PE events to see if they fulfil protocol definition.
Time Frame: Up to Week 52
Population: The ITT analysis set included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 583 | 575 | 563
weeks | 49.000 [40.000 to NA] — NA indicates that upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events during the 52 weeks treatment period. | 50.714 [37.571 to NA] — NA indicates that upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events during the 52 weeks treatment period. | 36.714 [31.143 to 41.429]
Statistical Analysis 1: Comparison: Brensocatib 10 mg vs Placebo; Estimate of Cox proportional hazard model=effect for treatment, sputum sample for Pseudomonas aeruginosa at screening and PE [<3 or ≥3] in last 12 months, stratification region and age group. Robust sandwich covariance estimator used; Test type: Superiority; p = 0.01, Cox proportional hazard — Adjusted p-value = 0.0200. The enhanced mixture-based gatekeeping procedure was used to control the overall type I error rate. Multiplicity adjusted p-value for the secondary endpoints were tested at two-sided alpha = 0.05; Hazard Ratio (HR) = 0.813, 95% CI 2-sided [0.695 to 0.952]
Statistical Analysis 2: Comparison: Brensocatib 25 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0182, Cox proportional hazard — Adjusted p-value = 0.0364. The enhanced mixture-based gatekeeping procedure was used to control the overall type I error rate. Multiplicity adjusted p-value for the secondary endpoints were tested at two-sided alpha = 0.05; Hazard Ratio (HR) = 0.825, 95% CI 2-sided [0.703 to 0.968]

3. Secondary Outcome: Responder Status for Exacerbation-Free Over the 52-Week Treatment Period
Description: Responder status was based on percentage of participants who were exacerbation free over 52-weeks of treatment period. Pulmonary exacerbation was defined as having 3 or more of the following symptoms for at least 48 hours resulting in a physician's decision to prescribe antibiotics: 1. Increased cough 2. Increased sputum volume or change in sputum consistency 3. Increased sputum purulence 4. Increased breathlessness and/or decreased exercise tolerance 5. Fatigue and/or malaise 6. Hemoptysis. A minimum of 14 days must have occurred between one exacerbation onset and the next. Any exacerbation that occurred less than 14 days from the prior exacerbation was not considered a new exacerbation. Independent adjudication committee of pulmonary physicians adjudicated reported PE events to see if they fulfill protocol definition. For discontinuation prior to Week 52 without having experienced a confirmed PE, responder status was imputed by multiple imputation.
Time Frame: Up to Week 52
Population: The ITT analysis set included all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 583 | 575 | 563
percentage of participants | 48.5 | 48.5 | 40.3
Statistical Analysis 1: Comparison: Brensocatib 10 mg vs Placebo; Missing responder status was imputed 100 times. Dataset was analyzed via logistic regression with treatment group, sputum P. aeruginosa status, prior PEs (<3/≥3), region, and age group as fixed effects. Results were then combined using Rubin's rules; Test type: Superiority; p = 0.0059, Logistic Regression — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.412, 95% CI 2-sided [1.105 to 1.806]
Statistical Analysis 2: Comparison: Brensocatib 25 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0074, Logistic Regression — [p-value comment as in outcome 2, analysis 2]; Odds Ratio (OR) = 1.4, 95% CI 2-sided [1.095 to 1.792]

4. Secondary Outcome: Change From Baseline at Week 52 in Postbronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: FEV1 was used to assess lung function and is the maximum amount of air that can be forced out in one second after first second after taking a forced expiration as measured by spirometer. Postbronchodilator FEV1 tests included spirometry tests performed referred to the spirometry performed within 30 minutes after administration of bronchodilator (4 puffs of salbutamol/albuterol, terbutaline or ipratropium). A positive change from baseline indicates an improvement in lung function. Baseline was the most recent non-missing assessment determined as best effort prior to the first dose of the investigational product.
Time Frame: Baseline, Week 52
Population: The ITT analysis set included all participants who were randomized. 'Overall number of participants analyzed' indicates the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: liter (L)
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 564 | 551 | 539
liter (L) | -0.050 (0.0093) | -0.024 (0.0099) | -0.062 (0.0094)
Statistical Analysis 1: Comparison: Brensocatib 10 mg vs Placebo; Analysis on linear repeated measure model=treatment visit, sputum sample for Pseudomonas aeruginosa at start, PE [<3 or ≥3] last 12 months, stratification region, age group (fixed effect) & baseline (covariate). Robust sandwich covariance estimator used; Test type: Superiority; p = 0.3841, Linear repeated measures model — Adjusted p-value = 0.3841. The enhanced mixture-based gatekeeping procedure was used to control the overall type I error rate. Multiplicity adjusted p-value was tested at two-sided alpha = 0.05; Difference in Least square (LS) Mean = 0.011, 95% CI 2-sided [-0.014 to 0.037], Standard Error of Mean 0.0132
Statistical Analysis 2: Comparison: Brensocatib 25 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0054, Linear repeated measures model — Adjusted p-value = 0.0364. The enhanced mixture-based gatekeeping procedure was used to control the overall type I error rate. Multiplicity adjusted p-value was tested at two-sided alpha = 0.05; Difference in LS Mean = 0.038, 95% CI 2-sided [0.011 to 0.065], Standard Error of Mean 0.0136

5. Secondary Outcome: Annualized Rate of Severe PEs
Description: Pulmonary exacerbation was defined as having 3 or more of the following symptoms for at least 48 hours resulting in a physician's decision to prescribe antibiotics: 1. Increased cough 2. Increased sputum volume or change in sputum consistency 3. Increased sputum purulence 4. Increased breathlessness and/or decreased exercise tolerance 5. Fatigue and/or malaise 6. Hemoptysis. A severe PE was defined as those requiring IV antibacterial drug treatment and/or hospitalization. A minimum of 14 days must have occurred between one exacerbation onset and the next. Any exacerbation that occurred less than 14 days from the prior exacerbation was not considered a new exacerbation. Independent adjudication committee with pulmonary physicians adjucated reported PE events to see if they fulfil the protocol definition. The rate of PE was analyzed using the negative binomial model.
Time Frame: Up to Week 52
Population: The ITT analysis set included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: exacerbation per participant-year
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 583 | 575 | 563
exacerbation per participant-year | 0.137 [0.103 to 0.182] | 0.137 [0.105 to 0.179] | 0.185 [0.142 to 0.242]
Statistical Analysis 1: Comparison: Brensocatib 10 mg vs Placebo; Analysis based on a negative binomial model including treatment, sputum sample for Pseudomonas aeruginosa at screening, PE [<3 or ≥3] in previous 12 months, stratification region and age group. Robust sandwich covariance estimator used; Test type: Superiority; p = 0.1277, Negative binomial regression — [p-value comment as in outcome 4, analysis 1]; Rate ratio = 0.742, 95% CI 2-sided [0.505 to 1.089]
Statistical Analysis 2: Comparison: Brensocatib 25 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1025, Negative binomial regression — Adjusted p-value = 0.2050. The enhanced mixture-based gatekeeping procedure was used to control the overall type I error rate. Multiplicity adjusted p-value was tested at two-sided alpha = 0.05; Rate ratio = 0.74, 95% CI 2-sided [0.515 to 1.062]

6. Secondary Outcome: Change From Baseline at Week 52 in Quality of Life Questionnaire - Bronchiectasis (QOL-B) Respiratory Symptoms Domain Score in Adult Participants
Description: The QOL-B is a validated, self-administered patient-reported outcome (PRO) that assesses symptoms, functioning, and health-related quality of life for participants with non-cystic fibrosis bronchiectasis (NCFBE). It contains 37 items in 8 domains (Respiratory Symptoms, Physical Functioning, Role Functioning, Emotional Functioning, Social Functioning, Vitality, Health Perceptions and Treatment Burden). Each of the 37 items is scored from 1 to 4, and each of the 8 domains scale scores is standardized on a 0-100 point scale, with higher scores representing fewer symptoms or better functioning. A positive change from Baseline indicates improvement in symptoms. For this outcome measure, change in the respiratory symptoms domain score from Baseline was reported. Baseline refers to most recent assessment on or before study Day 1.
Time Frame: Baseline, Week 52
Population: The ITT analysis set included all participants who were randomised. Overall number of participants analyzed indicates the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 487 | 495 | 486
score on scale | 6.841 (0.7706) | 8.575 (0.7556) | 4.809 (0.7500)
Statistical Analysis 1: Comparison: Brensocatib 10 mg vs Placebo; Analysis based on a linear repeated measures model with treatment group, visit, sputum sample for Pseudomonas aeruginosa at screening, pulmonary exacerbations [<3 or ≥3] in previous 12 months, stratification region fixed effect, baseline as covariate; Test type: Superiority; p = 0.0594, linear repeated measures model — [p-value comment as in outcome 4, analysis 1]; LS mean difference = 2.031, 95% CI 2-sided [-0.081 to 4.143], Standard Error of Mean 1.0775
Statistical Analysis 2: Comparison: Brensocatib 25 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0004, linear repeated measures model — [p-value comment as in outcome 5, analysis 2]; LS mean difference = 3.766, 95% CI 2-sided [1.680 to 5.852], Standard Error of Mean 1.0642

7. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs are AEs that occurred on or after the date of first dose of study drugs and within 28 days after the end of treatment.
Time Frame: Up to Week 56
Population: The Safety analysis set included all participants who were randomized and received at least 1 dose of brensocatib or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
Number analyzed (Participants) | 582 | 574 | 563
Participants | 452 | 440 | 448

8. Secondary Outcome: Plasma Concentration of Brensocatib in Adults (Main Study)
Time Frame: 2 hours (h) post-dose on Day 1; Pre-dose and 2 h post-dose at Weeks 4, 28 and 40; Pre-dose at Weeks 16 and 52
Population: The Pharmacokinetics (PK) concentration analysis set included adult participants who consented to participate in the main study in adult's cohort, received at least 1 dose of brensocatib, and had at least 1 postdose plasma concentration of brensocatib. 'Overall number of participants analyzed' indicates the number of participants with data available for analysis. 'Number analyzed' signifies number of adult participants with data available for analysis at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg
Number analyzed (Participants) | 194 | 208
nanograms per milliliter (ng/ml)
  Day 1: 2 h post-dose: number analyzed (Participants) | 18 | 24
  Day 1: 2 h post-dose | 40.52 (69.1) | 134.9 (51.4)
  Week 4: Pre-dose: number analyzed (Participants) | 56 | 63
  Week 4: Pre-dose | 52.60 (68.7) | 157.4 (70.8)
  Week 4: 2 h post-dose: number analyzed (Participants) | 20 | 25
  Week 4: 2 h post-dose | 100.5 (32.8) | 293.6 (35.1)
  Week 16: Pre-dose: number analyzed (Participants) | 94 | 105
  Week 16: Pre-dose | 45.19 (55.0) | 131.6 (69.0)
  Pre-dose at Week 28: number analyzed (Participants) | 120 | 130
  Pre-dose at Week 28 | 49.30 (63.9) | 143.0 (64.6)
  Week 28: 2 h post-dose: number analyzed (Participants) | 40 | 36
  Week 28: 2 h post-dose | 91.79 (45.3) | 323.7 (40.1)
  Week 40: Pre-dose: number analyzed (Participants) | 164 | 176
  Week 40: Pre-dose | 45.71 (54.2) | 136.8 (63.4)
  Week 40: 2 h post-dose: number analyzed (Participants) | 47 | 43
  Week 40: 2 h post-dose | 107.3 (45.0) | 302.6 (40.7)
  Week 52: Pre-dose | 45.78 (61.7) | 135.4 (60.3)

9. Secondary Outcome: Plasma Concentration of Brensocatib in Adults (PK Substudy)
Time Frame: 0.5 h, 2 h, and 4 to 8 h post-dose on Day 1and at Week 28; Pre-dose and 2 h post-dose at Weeks 4 and 48; Pre-dose at Weeks 16 and 52
Population: The PK concentration analysis set included adult participants who consented to participate in the PK substudy and received at least 1 dose of brensocatib, and had at least 1 postdose plasma concentration of brensocatib. 'Overall number of participants analyzed' indicates the number of participants with data available for analysis. 'Number analyzed' signifies number of adult participants with data available for analysis at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg
Number analyzed (Participants) | 62 | 64
ng/ml
  Day 1: 0.5 h post-dose | 34.51 (97.9) | 85.13 (103.5)
  Day 1: 2 h post-dose | 44.52 (55.0) | 120.0 (56.2)
  Day 1: 4-8 h post-dose: number analyzed (Participants) | 61 | 64
  Day 1: 4-8 h post-dose | 38.13 (52.9) | 108.5 (46.9)
  Week 4: Pre-dose: number analyzed (Participants) | 60 | 60
  Week 4: Pre-dose | 57.53 (53.4) | 131.3 (60.2)
  Week 4: 2 h post-dose: number analyzed (Participants) | 59 | 61
  Week 4: 2 h post-dose | 100.3 (44.1) | 286.7 (38.4)
  Week 16: Pre-dose: number analyzed (Participants) | 61 | 58
  Week 16: Pre-dose | 50.24 (58.1) | 138.0 (64.5)
  Week 28: Pre-dose: number analyzed (Participants) | 61 | 59
  Week 28: Pre-dose | 50.33 (54.7) | 124.6 (59.8)
  Week 28: 0.5 h post-dose: number analyzed (Participants) | 56 | 55
  Week 28: 0.5 h post-dose | 89.75 (46.0) | 235.5 (53.3)
  Week 28: 2 h post-dose: number analyzed (Participants) | 58 | 58
  Week 28: 2 h post-dose | 95.33 (35.3) | 271.9 (46.0)
  Week 28: 4-8 h post-dose: number analyzed (Participants) | 56 | 53
  Week 28: 4-8 h post-dose | 86.27 (40.7) | 246.4 (43.7)
  Week 40: Pre-dose: number analyzed (Participants) | 58 | 55
  Week 40: Pre-dose | 51.80 (54.4) | 119.3 (51.3)
  Week 40: 2 h post-dose: number analyzed (Participants) | 57 | 56
  Week 40: 2 h post-dose | 93.74 (32.1) | 271.2 (45.0)
  Week 52: Pre-dose: number analyzed (Participants) | 52 | 50
  Week 52: Pre-dose | 49.93 (72.2) | 131.6 (56.5)

10. Secondary Outcome: Plasma Concentration of Brensocatib in Adolescents (Main Study)
Time Frame: 0.5 h, 2 h, and 4 to 8 h post-dose on Day 1 and at Week 28; Pre-dose and 2 h post-dose at Weeks 4 and 48; Pre-dose at Weeks 16 and 52
Population: The PK concentration analysis set included adolescent participants who consented to participate in the main study and received at least 1 dose of brensocatib, and had at least 1 postdose plasma concentration of brensocatib. 'Overall number of participants analyzed' indicates the number of participants with data available for analysis. 'Number analyzed' signifies number of adolescent participants with data available for analysis at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg
Number analyzed (Participants) | 14 | 16
ng/ml
  Day 1: 0.5 h post-dose: number analyzed (Participants) | 12 | 14
  Day 1: 0.5 h post-dose | 63.20 (51.7) | 109.3 (139.1)
  Day 1: 2 h post-dose: number analyzed (Participants) | 13 | 14
  Day 1: 2 h post-dose | 68.33 (32.5) | 202.5 (50.7)
  Day 1: 4-8 h post-dose: number analyzed (Participants) | 12 | 14
  Day 1: 4-8 h post-dose | 56.07 (24.1) | 196.1 (52.4)
  Week 4: Pre-dose | 44.10 (64.2) | 126.6 (90.4)
  Week 4: 2 h post-dose: number analyzed (Participants) | 13 | 16
  Week 4: 2 h post-dose | 134.9 (52.8) | 432.9 (44.3)
  Week 16: Pre-dose: number analyzed (Participants) | 14 | 15
  Week 16: Pre-dose | 40.62 (51.6) | 158.1 (95.7)
  Week 28: Pre-dose: number analyzed (Participants) | 14 | 11
  Week 28: Pre-dose | 43.74 (57.2) | 132.9 (96.3)
  Week 28: 0.5 h post-dose: number analyzed (Participants) | 11 | 10
  Week 28: 0.5 h post-dose | 123.4 (49.1) | 321.6 (93.8)
  Week 28: 2 h post-dose: number analyzed (Participants) | 13 | 10
  Week 28: 2 h post-dose | 118.5 (30.5) | 336.9 (77.7)
  Week 28: 4-8 h post-dose: number analyzed (Participants) | 11 | 10
  Week 28: 4-8 h post-dose | 115.4 (27.7) | 309.9 (48.0)
  Week 40: Pre-dose: number analyzed (Participants) | 10 | 7
  Week 40: Pre-dose | 37.30 (52.5) | 84.39 (102.3)
  Week 40: 2 h post-dose: number analyzed (Participants) | 10 | 7
  Week 40: 2 h post-dose | 110.4 (43.9) | 262.8 (77.6)
  Week 52: Pre-dose: number analyzed (Participants) | 6 | 7
  Week 52: Pre-dose | 43.02 (64.8) | 104.0 (57.8)

ADVERSE EVENTS:
Time Frame: Up to Week 56
Description: The safety analysis set included all participants who were randomized and received at least 1 dose of brensocatib or placebo.
Arm/Group | Brensocatib 10 mg | Brensocatib 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/582 | 4/574 | 8/563
Serious Adverse Events (participants affected / at risk) | 101/582 | 97/574 | 108/563
Other Adverse Events (participants affected / at risk) | 197/582 | 213/574 | 203/563
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Brensocatib 10 mg (N=582) | Brensocatib 25 mg (N=574) | Placebo (N=563)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 4
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Blindness transient (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 3
Cataract nuclear (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1
Vitreoretinal traction syndrome (Eye disorders) | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Biliary cyst (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 1
Aspergillus infection (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Bronchitis fungal (Infections and infestations) | 1 | 0 | 0
Burkholderia gladioli infection (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 4 | 9 | 6
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Coronavirus infection (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis cryptosporidial (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 1
Influenza (Infections and infestations) | 2 | 1 | 1
Klebsiella infection (Infections and infestations) | 0 | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Lung abscess (Infections and infestations) | 0 | 2 | 1
Mastitis (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 11 | 13 | 16
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 2 | 2 | 2
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1
Scrub typhus (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body in throat (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1/573 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Urinary sediment abnormal (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0/562
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Device dislocation (Product Issues) | 1 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 0
Pelvic organ prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 47 | 48 | 67
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brensocatib 10 mg (N=582) | Brensocatib 25 mg (N=574) | Placebo (N=563)
COVID-19 (Infections and infestations) | 89 | 113 | 83
Nasopharyngitis (Infections and infestations) | 45 | 36 | 43
Urinary tract infection (Infections and infestations) | 27 | 30 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 17 | 35
Headache (Nervous system disorders) | 39 | 49 | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 35 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT04594369/Prot_002.pdf
  • Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT04594369/SAP_001.pdf